CLINICAL TRIAL: NCT03027856
Title: A Sirolimus Eluting Bioresorbable Magnesium Stent for Treatment of Coronary Bifurcation Lesions - The BIFSORB Pilot Study II
Brief Title: The BIFSORB Pilot Study II
Acronym: BIFSORB P-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, Principal investigator (MD, PhD), Aarhus University Hospital Skejby
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1-10-72-194-16
Record Dates: First submitted 2016-11-22; First posted 2017-01-23 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous intervention (PCI); Optical coherence tomography (OCT); Bifurcation lesion; Bioresorbable stents (BRS)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Magmaris (Experimental): Implantation of sirolimus eluting bioresorbable magnesium stent
  Interventions: Device: Magmaris

INTERVENTIONS:
Device: Magmaris — Implantation of a sirolimus eluting bioresorbable magnesium stent

SUMMARY:
The purpose of this study is to investigate the feasibility and safety of the Magmaris BRS for treatment of coronary bifurcation lesions.

DETAILED DESCRIPTION:
Bioresorbable stents are promising in treatment of coronary artery disease. The concept of bifurcation treatment using BRS is particular appealing as struts covering the side branch ostium may resorb over time.

The aim of this study is to investigate the feasibility and safety of the Magmaris BRS for treatment of coronary bifurcation lesions.

Hypothesis: treatment of coronary bifurcation lesions using the Magmaris BRS is safe and feasible.

Methods:

The study is a proof-of-concept, prospective, single arm study with inclusion of 20 patients. Planned 1-and 12-month follow-up by optical coherence tomography (OCT) and follow-up for clinical endpoints until 5 years.

Written informed consent is required before the procedure is performed. Eligible patients with a bifurcation lesion are treated by the provisional technique with mandatory jailing of the side branch and provisional opening of side branch ostium by the mini-kiss technique in case of severe pinching or TIMI-flow less than III. Proximal post-dilatation is mandatory. No dilatation beyond the expansion limits of the stent.

At baseline, the target lesion is assessed by OCT before, during and after implantation of the Magmaris BRS. OCT assessment is performed again at 1- and 12-month follow-up, or before if the patient is readmitted with a possible target lesion failure.

The operator is not blinded to the OCT images as pre-PCI images should be used for sizing and positioning of the stent, and procedural OCT images are used to optimize stent implantation before performing final OCT.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris
* Stabilized non-ST elevation myocardial infarction
* Silent angina pectoris
* Age > 18 years
* De novo coronary bifurcation lesion at LAD/diagonal, CX/obtuse marginal or RCA-PDA/posterolateral branch
* All Medina classes except Medina x.x.1.
* Diameter of side branch ≥ 2.5 mm
* Side branch diameter stenosis less than 50%
* Signed informed consent

Exclusion Criteria:

* ST-elevation infarction within 48 hours
* Expected survival < 1 year
* Severe heart failure (NYHA≥III)
* S-creatinine > 120 µmol/L or GFR < 0.45 mL/min per 1.73 m2
* Allergy to contrast media, aspirin, clopidogrel, ticagrelor, ticlopidine or sirolimus
* Unable to cover main vessel lesion with one stent
* Severe tortuosity
* Severe calcification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Combined endpoint of: major procedural myocardial infarction, non-procedural myocardial infarction, target lesion failure and cardiac death | 1 month
  Combined endpoint of: major procedural myocardial infarction, non-procedural myocardial infarction, target lesion failure and cardiac death
Index of adverse vessel wall features by OCT | 1 month
  Index based on: side branch ostial area late loss, strut fracture, uncovered non-side branch apposed stent struts, uncovered stent struts in front of side branch, uncovered stent struts on acquired or persistent malapposed struts, persistent malapposition, max neointimal thickness/area stenosis, cumulated extra stent lumen gain

SECONDARY OUTCOMES:
Optical coherence tomography endpoint: Acute malapposition | Baseline
Optical coherence tomography endpoint: Acquired malapposition | 1 month
Optical coherence tomography endpoint: Persistent malapposition | 1 month
Optical coherence tomography endpoint: Coverage of jailing struts | 1 month
Optical coherence tomography endpoint: Extra stent lumen (including evaginations) | Baseline and 1 month
Optical coherence tomography endpoint: Late stent recoil | 1 month
Optical coherence tomography endpoint: Stent fracture | Baseline and 1 month
Optical coherence tomography endpoint: Single end attached protruding (floating) struts or neointimal tissue resembling struts | Baseline and 1 month
Optical coherence tomography endpoint: Ostial strut loss | Baseline and 1 month
Optical coherence tomography endpoint: Mean neointimal thickness | 1 month
Optical coherence tomography endpoint: Stent strut coverage | 1 month
Optical coherence tomography endpoint: Minimal luminal area in segmental analysis | Baseline and 1 month
Optical coherence tomography endpoint: Minimal stent area in segmental analysis | Baseline and 1 month
Optical coherence tomography endpoint: Minimum stent expansion area % | Baseline and 1 month
Optical coherence tomography endpoint: Segmental area stenosis | Baseline and 1 month
Optical coherence tomography endpoint: Healing above calcified plaque | 1 month
Optical coherence tomography endpoint: Healing above lipid plaque | 1 month
Optical coherence tomography endpoint: Acute thrombus on struts | Baseline
Optical coherence tomography endpoint: Late thrombus on struts | 1 month
Optical coherence tomography endpoint: Acute expansion | Baseline
  Measured in segments with: 1) calcified plaque, 2) lipid plaque, 3) area after predilatation < 30% of reference area, 4) stenosed segments (>50% area stenosis) with no dissections after predilatation
Optical coherence tomography endpoint: Late recoil | 1 month
  Measured in segments with: 1) calcified plaque, 2) lipid plaque, 3) area after predilatation < 30% of reference area, 4) stenosed segments (>50% area stenosis) with no dissections after predilatation
Angiographic endpoint: Ostial side branch area stenosis | Baseline and 1 month
Angiographic endpoint: Ostial side branch acute gain after main vessel stenting | Baseline
Angiographic endpoint: Ostial side branch late loss | 1 month
Angiographic endpoint: Ostial distal main vessel area stenosis | Baseline and 1 month
Angiographic endpoint: Ostial distal main vessel acute gain after main vessel stenting | Baseline
Angiographic endpoint: Ostial distal main vessel late loss | 1 month
Angiographic endpoint: Proximal main vessel area stenosis | Baseline and 1 month
Angiographic endpoint: Proximal main vessel acute gain after main vessel stenting | Baseline
Angiographic endpoint: Proximal main vessel late loss | 1 month
Angiographic endpoint: Minimal luminal area of all segments | Baseline and 1 month
Procedural endpoint: Procedure time | Intraoperative
Procedural endpoint: Contrast use in mL | Intraoperative
Procedural endpoint: Fluoroscopy time | Intraoperative
Combined endpoint of: major procedural myocardial infarction, non-procedural myocardial infarction, target lesion failure and cardiac death | 6 months
  Combined endpoint of: major procedural myocardial infarction, non-procedural myocardial infarction, target lesion failure and cardiac death
Combined endpoint of: major procedural myocardial infarction, non-procedural myocardial infarction, target lesion failure and cardiac death | 24 months
  Combined endpoint of: major procedural myocardial infarction, non-procedural myocardial infarction, target lesion failure and cardiac death
Combined endpoint of: major procedural myocardial infarction, non-procedural myocardial infarction, target lesion failure and cardiac death | 60 months
  Combined endpoint of: major procedural myocardial infarction, non-procedural myocardial infarction, target lesion failure and cardiac death

OTHER OUTCOMES:
Clinical endpoint: myocardial infarction | 5 years
Clinical endpoint: target lesion failure | 5 years
Clinical endpoint: target lesion revascularization | 5 years
Clinical endpoint: stent thrombosis | 5 years
Clinical endpoint: cardiac death | 5 years
Clinical endpoint: non-cardiac death | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Evald H Christiansen, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided